CLINICAL TRIAL: NCT02124655
Title: Antiplaque Effect of Essential Oils and 0.2% Chlorhexidine on an in Situ Model of Oral Biofilm Growth: a Randomised Clinical Trial.
Brief Title: Antiplaque Effect of Essential Oils and 0.2% Chlorhexidine on an in Situ Model of Oral Biofilm Growth.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Inmaculada Tomas, Senior Lecturer, University of Santiago de Compostela
Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 393/2012
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Oral Biofilm; Mouthwash; Periodontitis
Keywords: Biofilms; Chlorhexidine; Microscopy, confocal; Dental plaque; Mouthwashes
MeSH Terms: conditions — Periodontitis; Dental Plaque | interventions — Oils, Volatile; Listerine; Chlorhexidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Essential oils/0.2% chlorhexidine/Sterile water (Experimental): A) 20 ml rinses for 30 seconds with essential oils/2 times daily (1/0/1). -----14 days----- B) 10 mL rinses for 30 seconds with 0.2% chlorhexidine/2 times daily (1/0/1). -----14 days----- C) 20 mL rinses for 30 seconds with sterile water (1/0/1).
  Interventions: Drug: Essential oils; Drug: 0.2% chlorhexidine; Drug: Sterile water

INTERVENTIONS:
Drug: Essential oils
  Other Names: Listerine
Drug: 0.2% chlorhexidine
  Other Names: Oraldine Perio
Drug: Sterile water

SUMMARY:
The accumulation and maturation of oral biofilm in the gingival margin is widely recognised to be the primary aetiological factor in the development of chronic gingivitis. Based on this association, the current treatment of gingivitis is focused on biofilm disruption, which will normally include mechanical processes, both professionally and at home. However, for patients, it is not easy to achieve a proper level of plaque control. The efficient plaque control techniques are very time consuming and require a special motivation and skills for their optimum use. It was at this point where mouthwashes become important, due to the fact that they include diverse types of antimicrobial agents to complement the results of mechanical oral hygiene measures.

Chlorhexidine is considered the "gold standard" of oral antiseptics; nevertheless it has not been recommended for long periods of time due to its well-known secondary effects. All of these inconveniences have limited its acceptability among dental professionals and users; in contrast, however, are the exceptional antiseptic properties, promoting the interest of researchers in other alternative antiplaque agents. Mouthwashes containing essential oils in their formulation have received a lot of attention. Their antiplaque activity has been demonstrated in numerous clinical studies, in which they were used in conjunction with mechanical oral hygiene measures.

In order to achieve a better understanding of the clinical effects that antimicrobial agents produce in the interior of the biofilm, it is necessary to apply a methodology in which the biofilm grows directly in the interior of the oral cavity but its three dimensional structure is not distorted by manipulation.

The aim of this study was to evaluate the in situ antiplaque effect of 2 antimicrobial agents (essential oils formulation and 0.2% chlorhexidine) in the short term with a posterior analysis on "non-destructured" biofilm with Confocal Laser Scanning Microscope combined with fluorescence staining.

DETAILED DESCRIPTION:
The volunteers wore two individualised splint which was capable of holding 6 glass disks (6 mm in diameter, 1 mm thickness); this was polished at 800 grit. . These splints are formed of 2 sheets, an internal 1 mm soft vinyl sheet where the disks are attached and an external 1 mm rigid one made of polyethylene terephtalate that is fenestrated.

• Mouthwash protocol During the 96 hour (4 days) duration of each course of study, each volunteer wore the splints with the glass disks, withdrawing them from the oral cavity only during meals (they were stored in an opaque container in humid conditions) and to perform oral hygiene procedures, using only the mechanical removal of bacterial plaque with water, without the use of any toothpaste or mouthwash.

Using the permitted mechanical oral hygiene measures (without the splints), the volunteers performed the following protocols based on the manufacturers' instructions, with the splints in the oral cavity, during the 4 days in the morning (8.30) after breakfast and at night (22.00) after dinner:

A) 20 ml rinses for 30 seconds with essential oils/2 times daily. ----14 days---- B) 10 mL rinses for 30 seconds with 0.2% chlorhexidine/2 times daily. ----14 days---- C) 20 mL rinses for 30 seconds with sterile water (negative control). Using an internet-based balanced randomisation system, indicating the mouthwash that each subject would use first, second and third, all volunteers performed the 3 rinsing cycles, with a rest period of 14 days between each test.

• Collection of the samples of Plaque like-biofilm Sample collection was done individually at 8 am in the morning, so that the samples of each volunteer were analysed on different days. It was determined that a minimum of 10 hours should have elapsed since the last mouthwash on the previous night.

As the glass disks were removed from the splint, they were immediately immersed in 100 µL of fluorescence solution LIVE/DEAD® BacLight™ and kept in a dark chamber at room temperature for 15 minutes. Microscopic observation was performed by a single investigator who was unaware of the study design, using a Leica TCS SP2 laser scanning spectral confocal microscope (Leica Microsystems Heidelberg GmbH, Mannheim, Germany) with an HCX APOL 63x/0.9 water-immersion lens.

• Processing of the samples of Plaque like-Biofilm Four selected fields or XYZ series in the central part of each disk were evaluated. These fields were considered representative of the whole sample after the observer's general examination. Fluorescence emission was determined in a series of XY images in which each image corresponded to each of the Z positions (depth). The optical sections were scanned in 1 µm sections from the surface of the biofilm to its base, measuring the maximum thickness of the field and subsequently the mean thickness of the biofilm of the corresponding sample. The maximum thickness of biofilm field was defined as the distance between the substrate (in perpendicular) and the peaks of the highest cell clusters. The maximum biofilm thickness of each field was divided into 3 zones or equivalent layers: outer layer (layer 1), middle layer (layer 2) and inner layer (layer 3).

The capture of the data was done with the same settings in all cases. The spatial scan mode (XYZ) and the 1024x1024 pixels scan format resolution were used. The Argon-ion and DPSS laser were used at a 13% and 78% of maximum intensity, respectively. The values for the pinhole, zoom and scan speed were 121.58 microns, 1 and 400Hz, respectively. The only values that were different depending on the sample were the offset (range between -1% to 1%) and PMT gain which was different for channel red and green, being in general terms, higher for green than for red (test and positive control), due to the fact that there was more presence of green than red signal, being for the negative control the opposite. These values were always adjusted to get a good quality capture without background noise, avoiding excessive saturation of the brightest pixels of the image. As the technician was blind to the experiment, they were advised to make the adjustments always consistent with what was seeing by the objective of the microscope, obtaining an image which was the closest as possible to reality.

Quantification of bacterial vitality in the series of XY images was determined using cytofluorographic analysis (Leica Confocal Software). In this analysis, the images of each fluorochrome were defined as "channels" (SYTO 9 occupies the green channel and propidium iodide the red channel). Square capture masks were used to measure the area occupied (µm2) by the pixels in each channel, determining the total area occupied by the biofilm and the corresponding percentage of vitality. The intensity ranges that were considered as positive signal were between 100 and 255. Determination of the mean percentage of bacterial vitality in each field required sections with a minimum area of biofilm of 250 µm2, and the mean percentage of bacterial vitality of the biofilm was calculated for the corresponding sample and for each biofilm layer.

For quantification of the percentage of surface substrate covered by the biofilm (covering grade), the cytofluorogram itself was used. From the maximum projection (superposition of all planes captured) of each of the analysed fields, the percentage of covering grade was obtained by calculating the sum of the bacterial mass (vital and non-vital) in regard to the total surface of the field (% positive within total area).

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy adults.
* Minimum of 24 permanent teeth.
* No gingivitis (Community Periodontal Index score = 0).
* No periodontitis (Community Periodontal Index score = 0).
* Absence of untreated caries.

Exclusion Criteria:

* Smoker or former smoker.
* Presence of dental prostheses.
* Presence of orthodontic devices.
* Antibiotic treatment or routine use of oral antiseptics in the previous 3 months.
* Presence of any systemic disease that could alter the production or composition of saliva.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Bacterial vitality (%) | 10 hours after the last mouthwash
  ratio of alive/dead bacteria.
Biofilm thickness (microns) | 10 hours after the last mouthwash
  thickness of the biofilm from the base of the substrate to the top surface of the biofilm
covering grade (%) | 10 hours after the last mouthwash
  area of the substrate that is covered by the biofilm after the 4 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Tomas, Principal Investigator — Senior lecturer at the University of Santiago de Compostela
Locations (1):
- Faculty of Medicine and Dentistry of the University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

REFERENCES:
- [Background] Garcia-Caballero L, Quintas V, Prada-Lopez I, Seoane J, Donos N, Tomas I. Chlorhexidine substantivity on salivary flora and plaque-like biofilm: an in situ model. PLoS One. 2013 Dec 27;8(12):e83522. doi: 10.1371/journal.pone.0083522. eCollection 2013. PMID 24386220
- [Background] Quintas V, Prada-Lopez I, Prados-Frutos JC, Tomas I. In situ antimicrobial activity on oral biofilm: essential oils vs. 0.2 % chlorhexidine. Clin Oral Investig. 2015 Jan;19(1):97-107. doi: 10.1007/s00784-014-1224-3. Epub 2014 Apr 1. PMID 24687247
- [Derived] Quintas V, Prada-Lopez I, Donos N, Suarez-Quintanilla D, Tomas I. Antiplaque effect of essential oils and 0.2% chlorhexidine on an in situ model of oral biofilm growth: a randomised clinical trial. PLoS One. 2015 Feb 17;10(2):e0117177. doi: 10.1371/journal.pone.0117177. eCollection 2015. PMID 25689859